CLINICAL TRIAL: NCT07022236
Title: Assessment of Thyroid Dysfunction in Patients Undergoing Haemodialysis at Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Elsayed, Internal Medicine Resident, Sohag University
Other Study IDs: Soh-Med--25-4-012MS
Record Dates: First submitted 2025-05-24; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Dialysis; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thyroid profile — Thyroid dysfunction in patients undergoing hemogdialysis in sohag university hospital

SUMMARY:
Thyroid dysfunction is a prevalent endocrine disorder that significantly impacts the health of patients with chronic kidney disease (CKD), particularly those undergoing dialysis. The prevalence of thyroid dysfunction in dialysis patients has been reported to range from 20% to 60%, highlighting the need for routine screening and management in this vulnerable group (Kuo et al., 2024). Thyroid hormones play a crucial role in regulating various physiological processes, and their dysregulation can lead to complications such as cardiovascular disease, anemia, and impaired quality of life, which are particularly concerning in the dialysis population (Smith et al., 2024).

The relationship between CKD and thyroid dysfunction is complex and multifactorial. Uremic toxins can interfere with the hypothalamic-pituitary-thyroid axis, leading to alterations in thyroid hormone production and metabolism. Recent studies have shown that inflammation and oxidative stress associated with CKD can further exacerbate thyroid dysfunction (Johnson et al., 2024). Understanding these mechanisms is essential for developing effective management strategies for thyroid health in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Patients diagnosed with end-stage renal disease (ESRD) on regular hemodialysis for at least 3 months.

Exclusion Criteria:

* Known Thyroid Disorders: Patients with a history of thyroid disease (e.g., hypothyroidism, hyperthyroidism) prior to starting dialysis.
* Recent Thyroid Treatment: Patients who have received treatment for thyroid dysfunction (e.g., thyroid hormone replacement, antithyroid medications) within the last six months.
* Patients with acute kidney injury (AKI) or those who are not on regular dialysis.
* Pregnant or lactating women.
* Patients with systemic illnesses or medications that could interfere with thyroid function tests (e.g., corticosteroids, lithium).

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing hemodialysis in sohag university hospital
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Thyroid Dysfunction Diagnosed by Serum TSH, Free T3, and Free T4 Levels | Up to 6 months from enrollment
  Diagnosis will be classified as:
  Hypothyroidism Subclinical hypothyroidism Hyperthyroidism

SECONDARY OUTCOMES:
Number of Participants With Thyroid Dysfunction Stratified by Dialysis Duration and Ultrafiltration Rate | Up to 6 months from enrollment
  Number of Participants With Thyroid Dysfunction Stratified by Dialysis Duration and Ultrafiltration Rate Dialysis duration recorded in months Ultrafiltration rate recorded in mL/kg/hour Thyroid dysfunction diagnosed by TSH, free T3, and free T4 levels

OTHER OUTCOMES:
Number of Participants With Thyroid Dysfunction by Underlying Cause of Kidney Disease | Up to 6 months from enrollment
  Number of Participants With Thyroid Dysfunction by Underlying Cause of Kidney Disease
  Kidney disease categories:
  Diabetic nephropathy Hypertensive nephrosclerosis Chronic glomerulonephritis Thyroid dysfunction diagnosed by serum TSH, free T3, and free T4

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital, Sohag, Egypt